CLINICAL TRIAL: NCT01594697
Title: Metformin in Pregnancy in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Maurizio Guido, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000082011
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

ARMS (1):
- metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
The study provide a detailed longitudinal evaluation of the gluco-insulinemic assessment of pregnant PCOS women under metformin treatment. 47 non diabetic Polycystic Ovary Syndrome (PCOS) women became pregnant during metformin treatment and continued taking the drug during gestation. An oral glucose tolerance test and euglycaemic hyperinsulinaemic clamp were performed at each trimester of gestation.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 yr,
* metformin treatment for at least 3 months before entering the pregnancy,
* gestational age between 5 and 12 wk

Exclusion Criteria:

* diabetes mellitus
* significant liver or renal impairment
* neoplasms and other endocrine diseases
* the use of drugs other than metformin able to interfere with glucose and insulin metabolism.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Enrollment: 60 (Actual)

PRIMARY OUTCOMES:
incidence of gestational diabetes

SECONDARY OUTCOMES:
rate of spontaneous abortion
number of hypertensive disorders
number of live births
number of newborns with macrosomia
incidence of delivery by caesarian section

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Rome, Italy

REFERENCES:
- [Derived] Romualdi D, De Cicco S, Gagliano D, Busacca M, Campagna G, Lanzone A, Guido M. How metformin acts in PCOS pregnant women: insights into insulin secretion and peripheral action at each trimester of gestation. Diabetes Care. 2013 Jun;36(6):1477-82. doi: 10.2337/dc12-2071. Epub 2013 Jan 11. PMID 23315599